CLINICAL TRIAL: NCT05751239
Title: Motives for Desiring Children in Different Sexual-romantic Orientations: A Cross-sectional Study
Brief Title: Motives for Desiring Children in Different Sexual-romantic Orientations
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: BASEC 201800535
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Family Characteristics; Sexual Orientation
Keywords: Romantic orientation; Queer; Parenting
MeSH Terms: conditions — Sexual Behavior; Homosexuality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Bisexual-Biromantic: People that self-identify as bisexual-biromantic
  Interventions: Other: Questionaire
- Heterosexual-heteroromantic: People that self-identify as heterosexual-heteroromantic
  Interventions: Other: Questionaire
- Homosexual-homoromantic: People that self-identify as homosexual-homoromantic
  Interventions: Other: Questionaire
- Pansexual-panromantic: People that self-identify as pansexual-panromantic
  Interventions: Other: Questionaire

INTERVENTIONS:
Other: Questionaire — All participants answered an online questionaire. Out of the 837 participants 641 were included

SUMMARY:
The goal of this cross-sectional study is to compare the motives for the desire to have children in different sexual-romantic orientation. The main question[s] it aims to answer are:

* Do all orientations have the same motives for the desire to have children?
* What are the preferred methods for having a child for the different orientations

Participants will answer an online questionaire .

Researchers will compare the different orientations to see if there are differences.

ELIGIBILITY:
Inclusion Criteria:

* All participants regardless of sex, gender or age

Exclusion Criteria:

* Incomplete questionnaire
* Under 18 years
* Caring for a child in a social, economic or educational way (self-report)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: LGBT+ organisations and groups in Switzerland and social media were contacted for the participants' recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 837 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Possible difference in the motive to have a child between different orientations. | At baseline in July/August 2018
  The questionnaire, that was answered at baseline, included statements that people rated. There were 5 statement each for each motive and 10 additional statements

SECONDARY OUTCOMES:
Preferred way to have a child of the different orientations | At baseline in July/August 2018
  People with positive wish for child could choose from different possibilities their preferred method (assessed via questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Petra Stute, Dr. med., Study Chair — Department of Obstetrics and Gynecology, lnselspital, Bern University Hospital, University of Bern
Locations (1):
- Department of Obstetrics and Gynecology, lnselspital, Bern University Hospital, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No